CLINICAL TRIAL: NCT06608498
Title: User-Centered Design of a Single-Module Digital Mental Health Intervention for College Students at Risk for Psychosis
Brief Title: DMHI for At-Risk College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Buck, Assistant Professor; Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019663; P50MH115837 (NIH)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prodromal Symptoms; Psychosis
Keywords: College student mental health
MeSH Terms: conditions — Prodromal Symptoms; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (SPARK Coping) (Active Comparator): Participants will be given a link to SPARK Coping immediately following their baseline assessments are complete.
  Interventions: Behavioral: SPARK Coping
- Waitlist Control (No Intervention): Participants will wait until their follow-up assessment to be given access to the SPARK Coping intervention.

INTERVENTIONS:
Behavioral: SPARK Coping — SPARK Coping is a single-session intervention providing psychoeducation and structured practices related to stigma reduction, cognitive restructuring, behavioral activation, and effective coping. It is a self-guided website powered by research data capture software.
  Arms: Intervention (SPARK Coping)

SUMMARY:
The goal of this clinical trial is to learn if a single-session digital intervention (SPARK Coping) is acceptable, usable, and demonstrates a preliminary signal of efficacy in reducing symptom-related distress and increasing positive treatment-seeking attitudes among college students reporting subthreshold symptoms associated with risk for psychosis. Research questions inclue:

* Does SPARK Coping reduce symptom-related distress and increase positive treatment seeking attitudes (primary outcomes) relative to a waitlist control condition?
* Does SPARK Coping increase adaptive coping and reduce internalized stigma (primary targets) relative to a waitlist control condition?

Researchers will compare provision of SPARK Coping to a waitlist control condition and collect data from participants on each of the variables described above. Participants will:

* Complete questionnaires and surveys remotely at the start of the study and two weeks later
* Be offered access to the SPARK Coping intervention either after completion of their baseline assessment (intervention arm) or after two weeks (waitlist control arm).

ELIGIBILITY:
Inclusion Criteria:

* Symptoms indicating risk for psychosis (a distress score >= 20 on the Prodromal Questionnaire, Brief [PQ-B], per Savill et al., 2018; Early Intervention in Psychiatry and a positive frequency average score >= 1.47 on the Community Assessment of Psychic Experiences (CAPE-P15), per Jaya et al., 2021 and Bukenaite et al., 2017)
* Residence in the United States
* Currently enrolled in a post-secondary college program at the University of Washington.

Exclusion Criteria:

* Inconsistent or implausible reporting of symptoms at screening as determined by empirically-determined methods for detecting malingering or inconsistency
* Failure to demonstrate understanding of study details in comprehension screening

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Change in coping self-efficacy | Baseline, 2 weeks
  Caregiver coping self-efficacy will be assessed with the Coping Self-Efficacy Scale, a 26-item self-report questionnaire measuring the perceived ability of coping with various life challenges. Responses are rated on a 0 to 10 scale, and scores range from 0 to 260, with higher scores denoting a greater sense of self-efficacy in coping.
Change in internalized stigma | Baseline, 2 weeks
  Internalized stigma will be assessed with the Internalized Stigma of Mental Health Inventory, Brief (ISMI-9). The ISMI-9 is a nine-item self-report short form, where each item is rated on a four-point Likert scale (1 = Strongly disagree, 4 = Strongly agree), and higher scores indicate more severe internalization of mental illness stigma.
Change in attitudes toward treatment | Baseline, 2 weeks
  Help-Seeking Attitudes will be measured using the treatment and treatment-seeking subscales of the Endorsed and Anticipated Stigma Inventory (EASI). The full EASI is a 40-item self-reported questionnaire with subscales measuring beliefs about mental illness, beliefs about mental health treatment, beliefs about mental health treatment seeking, concerns about stigma from loved ones, and concerns about stigma from the workplace. The subscales are scored by summing the ratings from the eight individual items in each subscale (5-point scale with 1 = Strongly disagree, 5 = Strongly agree), with lower scores indicating less stigma, and more positive attitudes towards treatment and treatment-seeking. We will assess attitudes toward treatment and treatment-seeking by administering those two subscales. Total scores combining these two scales range from 16 to 80.
Change in positive psychosis symptom frequency and distress | Baseline, 2 weeks
  Distress related to positive psychosis symptoms will be assessed with the CAPE-P15, a 15-item measure of positive symptoms of psychosis and psychosis risk as well as distress associated with such experiences. These 15 items are rated both on frequency (1 = Never to 4 = Nearly always) and distress (1 = Not distressed to 4 = Very distressed).

SECONDARY OUTCOMES:
Change in recovery | Baseline, 2 weeks
  Recovery will be assessed using the Choice of Outcome in CBT for Psychoses, Short Form (CHOICE-SF). The CHOICE-SF is an 11-item self-report form developed to assess recovery-related goals for therapy. Participants rate themselves in different therapy-focused areas such as "self-confidence" or "ways of dealing with everyday stress" on a scale (0 = Worst, 10 = Best).
Change in general psychopathology / distress | Baseline, 2 weeks
  General psychopathology / distress will be assessed with General Health Questionnaire (GHQ), a 12-item questionnaire assessing general psychological morbidity. Respondents indicate agreement on a four-point scale (0 = Not at all; 3 = More than usual) and total scores ranging from 0 to 36 with higher scores indicating more severe psychological morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Buck, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States